CLINICAL TRIAL: NCT01226121
Title: A Post Market, Open-Label Study of the Safety and Efficacy of Delayed Manipulation After Xiaflex Treatment in Subjects With Dupuytren's Contracture
Brief Title: Safety and Efficacy of Delayed Manipulation After Xiaflex Treatment in Subjects With Dupuytren's Contracture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty enrolling additional patients
Sponsor: Indiana Hand to Shoulder Center (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: Principal Investigator, F. Thomas D. Kaplan, MD, MD, Indiana Hand to Shoulder Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHtSC-Delay 101
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Dupuytren's Disease
Keywords: dupuytren; dupuytren's
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Day 1 manipulation (Active Comparator): Finger manipulation one day following Clostridial collagenase injectable
  Interventions: Biological: Clostridial collagenase injectable
- Day 2 manipulation (Active Comparator): Finger manipulation two days following Clostridial collagenase injectable
  Interventions: Biological: Clostridial collagenase injectable
- Day 4 manipulation (Active Comparator): Finger manipulation four days following Clostridial collagenase injectable
  Interventions: Biological: Clostridial collagenase injectable

INTERVENTIONS:
Biological: Clostridial collagenase injectable — Finger manipulation performed 1, 2, or 4 days following collagenase injection

SUMMARY:
The purpose of this study is to determine if of manipulation of digits following collagenase injection for treatment of Dupuytren's contracture is effected by the amount of time between injection and manipulation.

DETAILED DESCRIPTION:
Patients with Metacarpophalangeal joint contractures caused by Dupuytren's disease will be evaluated as to the timing of the finger manipulation procedure that is performed following collagenase injection. Three groups will be evaluated: group 1 will have the manipulation procedure on the day following collagenase injection, group 2 will have the manipulation procedure on the second day following collagenase injection,and group 3 will have the manipulation procedure on the fourth day following collagenase injection,

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 18 years) of either gender with an metacarpophalangeal joint contracture and a palpable cord of > 20 degrees of a digit (excluding the thumb) due to Dupuytren's contracture

Exclusion Criteria:

* Any subject who has had prior surgical, percutaneous needle aponeurotomy or Xiaflex treatment for Dupuytren's contracture.
* Any subject using anti-coagulant therapy other than low dose aspirin (up to 150mg/day).
* Any subject in the opinion of the MD investigators with chronic, severe or terminal medical illness which would make them unsuitable for study participation.
* Any subject with known allergy to Xiaflex (Clostridial collagenase).
* Any subject who cannot conform to the study visit schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Thomas D. Kaplan, MD, Principal Investigator — Indiana Hand to Shoulder Center; Lawrence C Hurst, MD, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - Indiana Hand to Shoulder Center, Indianaplis, Indiana
  - Stony Brook University, Stony Brook, New York

REFERENCES:
- [Background] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771

RESULTS

PARTICIPANT FLOW:
Groups:
- Day 1 Manipulation: Finger manipulation one day following collagenase injection
- Day 2 Manipulation: Finger manipulation two days following collagenase injection
- Day 4 Manipulation: Finger manipulation four days following collagenase injection
Period: Overall Study
Arm/Group | Day 1 Manipulation | Day 2 Manipulation | Day 4 Manipulation
Started | 13 | 11 | 13
30 Day Evaluation | 12 | 11 | 13
Completed | 11 | 11 | 12
Not Completed | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Day 1 Manipulation | Day 2 Manipulation | Day 4 Manipulation | Total
Number analyzed (Participants) | 13 | 11 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.3) | 67 (6.4) | 65.5 (10.2) | 65.44 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 13 | 9 | 12 | 34
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clinical Improvement (> 50% Reduction in Contracture)
Time Frame: 30 days after injection
Measure: Number; unit: percentage of participants
Arm/Group | Day 1 Manipulation | Day 2 Manipulation | Day 4 Manipulation
Number analyzed (Participants) | 12 | 11 | 13
percentage of participants | 92 | 91 | 85

2. Secondary Outcome: Percentage of Patients Obtaining Clinical Success at 90 Days (<=5 Degree Residual Contracture)
Time Frame: 90 days
Measure: Number; unit: percentage of patients
Arm/Group | Day 1 Manipulation | Day 2 Manipulation | Day 4 Manipulation
Number analyzed (Participants) | 11 | 11 | 12
percentage of patients | 91 | 82 | 83

ADVERSE EVENTS:
Time Frame: data collected for 90 day period patients were followed following injection
Arm/Group | Day 1 Manipulation | Day 2 Manipulation | Day 4 Manipulation
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 11/11 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Day 1 Manipulation (N=13) | Day 2 Manipulation (N=11) | Day 4 Manipulation (N=13)
Edema (Skin and subcutaneous tissue disorders) | 13 | 9 | 10
Bruising (Skin and subcutaneous tissue disorders) | 9 | 8 | 9
Pain (Nervous system disorders) | 1 | 5 | 5
Blister (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2 | 0
Skin tear (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
pruritis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No